CLINICAL TRIAL: NCT03582813
Title: Randomized Controlled Trial of Mental Health Self-Directed Care Financing in Texas
Brief Title: Efficacy of Mental Health Self-Directed Care Financing
Acronym: SDC-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith A. Cook, Professor of Psychiatry, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0970; H133B050003 (Other Grant/Funding Number: US Dept of Educ-NIDRR Center for Mental Health Services Cooperative Agreement)
Record Dates: First submitted 2018-05-21; First posted 2018-07-11 (Actual); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Mental Illness Persistent
Keywords: self-directed care; mental health services; mental health recovery; behavioral health service financing

STUDY DESIGN:
Intervention Model Description: Self-directed care is a model of service delivery in which service recipients are allocated a individual budget from which they purchase mental health and other services and material goods needed to help them recover from their mental illness and remain outside of restrictive settings such as hospitals..
Who Masked: Outcomes Assessor
Masking Description: Research interviewers were blinded to study condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-directed care (Experimental): Subjects receive traditional behavioral health and non-traditional services via a self-directed care model in which they develop a person-directed plan and create a budget for the purchase of medically necessary goods and services. Program staff acting as service brokers help them secure needed goods and services from within or outside the public behavioral health provider system. A fiscal intermediary manages financial resources to pay providers and enable the purchase of approved goods..
  Interventions: Behavioral: Self-directed care
- Services as usual (Active Comparator): Subjects receive traditional behavioral health services as usual via the traditional service delivery system and its network of providers.
  Interventions: Behavioral: Services as usual

INTERVENTIONS:
Behavioral: Self-directed care — Traditional and non-traditional behavioral health services are chosen from within and outside the public mental health system
  Arms: Self-directed care
Behavioral: Services as usual — Traditional behavioral health services are chosen from along those delivered at the patient's community mental health agency
  Arms: Services as usual

SUMMARY:
Self-directed care (SDC) programs give people with disabilities control over public funds to purchase traditional behavioral health and non-traditional services in order to remain outside of institutional settings. The purpose of this study is to determine the effects of this model on participant outcomes, service costs, and user satisfaction among people with serious mental illness.

DETAILED DESCRIPTION:
Self-directed care (SDC) programs give people with disabilities control over public funds to purchase traditional behavioral health and non-traditional services in order to remain outside of institutional settings. The purpose of this study is to determine the effects of this model on participant outcomes, service costs, and user satisfaction among people with serious mental illness. Adults with serious mental illness served in the Texas public health system will be randomly assigned to SDC versus services as usual and assessed at baseline, 12-month, and 24-month follow-up. Mixed effects random-regression analysis will test for longitudinal changes in outcomes between the two study conditions. Differences in service costs will be analyzed using generalized linear models with negative binomial and zero-inflated negative binomial distribution. Non-traditional expenditures by the SDC participants will be examined descriptively. Service satisfaction in both study conditions will be assessed at one- and two-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* receiving mental health services at a Texas Department of State Health Services-funded mental health program
* diagnosis of serious mental illness consistent with federal Public Law 102-32
* assigned to a level of care eligible for a package of comprehensive clinical and rehabilitation services known as Service Package 3
* 18 years or older
* able to understand spoken English.

Exclusion Criteria:

* cognitive impairment
* homeless at time of recruitment
* history of violent behavior resulting in arrest and conviction in the past 10 years
* active substance use in the absence of substance use treatment
* enrollment in Medicare or dual beneficiary
* finances controlled by a third party (e.g., representative payee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Cook, PhD, Principal Investigator — University of Illinois at Chicago, Department of Psychiatry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scanlan JN, Hancock N, Honey A. The Recovery Assessment Scale - Domains and Stages (RAS-DS): Sensitivity to change over time and convergent validity with level of unmet need. Psychiatry Res. 2018 Mar;261:560-564. doi: 10.1016/j.psychres.2018.01.042. PMID 29407723
- [Background] Davis C, Kellett S, Beail N. Utility of the Rosenberg self-esteem scale. Am J Intellect Dev Disabil. 2009 May;114(3):172-8. doi: 10.1352/1944-7558-114.3.172. PMID 19374464
- [Background] Pearlin LI, Schooler C. The structure of coping. J Health Soc Behav. 1978 Mar;19(1):2-21. No abstract available. PMID 649936
- [Background] Williams GC, Deci EL. Internalization of biopsychosocial values by medical students: a test of self-determination theory. J Pers Soc Psychol. 1996 Apr;70(4):767-79. doi: 10.1037//0022-3514.70.4.767. PMID 8636897
- [Result] Cook JA, Shore S, Burke-Miller JK, Jonikas JA, Hamilton M, Ruckdeschel B, Norris W, Markowitz AF, Ferrara M, Bhaumik D. Mental Health Self-Directed Care Financing: Efficacy in Improving Outcomes and Controlling Costs for Adults With Serious Mental Illness. Psychiatr Serv. 2019 Mar 1;70(3):191-201. doi: 10.1176/appi.ps.201800337. Epub 2019 Jan 11. PMID 30630401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants ( who were active Texas Department of State Health Services (DSHS) were recruited at community mental health agencies by local research staff between March 2009 and September 2010.
Period: Overall Study
Arm/Group | Self-directed Care | Services as Usual
Started | 114 | 102
Completed | 95 | 81
Not Completed | 19 | 21
Not completed — Lost to Follow-up | 18 | 21
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-directed Care | Services as Usual | Total
Number analyzed (Participants) | 114 | 102 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (10.0) | 41.6 (9.5) | 41.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 58 | 134
  Male | 38 | 44 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 11 | 33
  Not Hispanic or Latino | 92 | 91 | 183
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 52 | 103
  White | 60 | 47 | 107
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
High school diploma/General Equivalency Degree [Count of Participants; unit: Participants] | 76 | 66 | 142
Diagnosis Category [Count of Participants; unit: Participants]
  Schizophrenia | 38 | 35 | 73
  Major Depressive Disorder | 43 | 45 | 88
  Bipolar I or II Disorder | 33 | 22 | 55
  Co-Occurring Substance Abuse | 20 | 17 | 37
Mental Health services cost in year prior to study [Mean (Standard Deviation); unit: Dollar Amount] | 4,390 (3.29) | 3,996 (3.83) | 4,204 (3.55)

OUTCOME MEASURES:

1. Primary Outcome: Recovery From Mental Illness
Description: This outcome is measured by the Recovery Assessment Scale (RAS). Recovery is a psychosocial outcome assessed via patient self-ratings on a 41-item scale using a 5-point Likert-Response format ranging from "strongly disagree" to "strongly agree". The minimum value for the RAS is 41 and the maximum is 205, with higher scores indicating a better outcome. Dimensions of recovery include personal confidence and hope, willingness to ask for help, goal and success orientation, reliance on others, and not being dominated by one's residual psychiatric symptoms.
Time Frame: Study entry (pre-intervention), 12 months later (midpoint of intervention), & 24 months later (end of intervention)
Population: The number reflected in the "Overall Number of Participants Analyzed" pertains to the number of participants who completed the baseline interview.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed Care | Services as Usual
Number analyzed (Participants) | 114 | 102
score on a scale
  T1 - Baseline (pre-intervention) | 148.0 (20.45) | 152.81 (22.21)
  T2 - 12 months later (intervention mid-point): number analyzed (Participants) | 94 | 77
  T2 - 12 months later (intervention mid-point) | 151.88 (21.77) | 154.56 (20.03)
  T3 - 24 months later (end of intervention): number analyzed (Participants) | 94 | 75
  T3 - 24 months later (end of intervention) | 152.17 (21.18) | 153.62 (22.02)
Statistical Analysis 1: Comparison: Self-directed Care vs Services as Usual; This mixed effects random regression analysis tested whether intervention participants would report larger increases than controls in self-perceived Recovery and that this effect would be maintained overtime;; Test type: Superiority; p < .01, Mixed Effects Random Regression; MIXREG Estimate = 4.27, Standard Error of Mean 1.61

2. Secondary Outcome: Change in Self-esteem
Description: Feelings of self-worth and confidence in general abilities as measured by the Rosenberg Self-Esteem Scale . Higher vales equal better self=esteem. Minimum = 10 and maximum = 40.
Time Frame: Study entry (pre-intervention), 12 months later (midpoint of intervention), & 24 months later (end of intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed Care | Services as Usual
Number analyzed (Participants) | 114 | 102
score on a scale
  T1 - Baseline (pre-intervention) | 23.97 (5.78) | 24.57 (5.49)
  T2 - 12 months later (intervention mid-point): number analyzed (Participants) | 99 | 81
  T2 - 12 months later (intervention mid-point) | 25.74 (5.64) | 25.74 (5.53)
  T3 - 24 months later (end of intervention): number analyzed (Participants) | 94 | 81
  T3 - 24 months later (end of intervention) | 25.42 (5.75) | 25.19 (5.59)
Statistical Analysis 1: Comparison: Self-directed Care vs Services as Usual; This mixed effects random regression analysis tested whether intervention participants would report larger increases than controls in self-esteem that would be maintained longitudinally; Test type: Superiority; p = .031, Mixed Effects Random Regression; MIXREG Estimate = .90, Standard Error of Mean 0.42

3. Secondary Outcome: Coping Mastery
Description: Change in subjects' sense of personal control over important life outcomes as measured by the Coping Mastery Scale. Higher values equal better coping mastery. Minimum = 2 and maximum = 49.
Time Frame: Study entry (pre-intervention), 12 months later (midpoint of intervention), & 24 months later (end of intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed Care | Services as Usual
Number analyzed (Participants) | 114 | 102
score on a scale
  T1 - Baseline (pre-intervention) | 2.60 (0.50) | 2.66 (0.46)
  T2 - 12 months later (intervention mid-point): number analyzed (Participants) | 99 | 81
  T2 - 12 months later (intervention mid-point) | 2.67 (0.52) | 2.69 (0.61)
  T3 - 24 months later (end of intervention): number analyzed (Participants) | 94 | 81
  T3 - 24 months later (end of intervention) | 2.79 (0.51) | 2.60 (0.60)
Statistical Analysis 1: Comparison: Self-directed Care vs Services as Usual; This mixed effects random regression analysis tested whether intervention participants would report larger increases than controls in coping mastery that would be maintained longitudinally; Test type: Superiority; p < 0.01, Mixed Effects Random Regression; MIXREG Estimate = 0.12, Standard Error of Mean 0.04

4. Secondary Outcome: Perceived Autonomy Support
Description: Perceived support for autonomously motivated change measured by the Learning Climate Questionnaire of Williams & Deci. Measures change in perception that service environment is supportive of autonomy to make decisions and choices. Higher score equals better autonomy support. Minimum = 4 and maximum = 105.
Time Frame: Study entry (pre-intervention), 12 months later (midpoint of intervention), & 24 months later (end of intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed Care | Services as Usual
Number analyzed (Participants) | 114 | 102
score on a scale
  T1 - Baseline (pre-intervention) | 4.74 (1.72) | 4.65 (1.82)
  T2 - 12 months later (intervention mid-point): number analyzed (Participants) | 98 | 81
  T2 - 12 months later (intervention mid-point) | 5.56 (1.33) | 4.85 (1.57)
  T3 - 24 months later (end of intervention): number analyzed (Participants) | 94 | 81
  T3 - 24 months later (end of intervention) | 5.44 (1.54) | 4.83 (1.84)
Statistical Analysis 1: Comparison: Self-directed Care vs Services as Usual; This mixed effects random regression analysis tested whether intervention participants would report larger increases than controls in perceived autonomy support that would be maintained longitudinally; Test type: Superiority; p = 0.030, Mixed Effects Random Regression; MIXREG Estimate = 0.29, Standard Error of Mean 0.13

5. Secondary Outcome: Number of Participants With Employment
Description: Change in employment status as measured by Bureau of Labor Statistics definition of paid employment: with paid employment versus without paid employment. Higher value equals with paid employment.
  Minimum = 0 and maximum = 1.
Time Frame: Study entry (pre-intervention), 12 months later (midpoint of intervention), & 24 months later (end of intervention)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Self-directed Care | Services as Usual
Number analyzed (Participants) | 114 | 102
Participants
  T1 - Baseline (pre-intervention) | 16 | 13
  T2 - 12 months later (intervention mid-point): number analyzed (Participants) | 99 | 78
  T2 - 12 months later (intervention mid-point) | 18 | 6
  T3 - 24 months later (end of intervention): number analyzed (Participants) | 94 | 81
  T3 - 24 months later (end of intervention) | 19 | 6
Statistical Analysis 1: Comparison: Self-directed Care vs Services as Usual; This mixed effects random regression analysis tested whether intervention participants would report greater likelihood of employment that would be maintained longitudinally; Test type: Superiority; p = 0.046, Regression, Logistic; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.01 to 4.74]

6. Secondary Outcome: Number of Participants Enrolled in Classes
Description: Change in education participation status as measured by U.S. Department of Education's definition of school enrollment: enrolled in classes requiring registration and fee payment versus not enrolled in classes. Higher value = enrolled in classes. Minimum = 0 and maximum = 1.
Time Frame: Study entry (pre-intervention), 12 months later (midpoint of intervention), & 24 months later (end of intervention)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Self-directed Care | Services as Usual
Number analyzed (Participants) | 114 | 102
Participants
  T1 - Baseline (pre-intervention) | 7 | 10
  T2 - 12 months later (intervention mid-point): number analyzed (Participants) | 99 | 78
  T2 - 12 months later (intervention mid-point) | 5 | 5
  T3 - 24 months later (end of intervention): number analyzed (Participants) | 94 | 81
  T3 - 24 months later (end of intervention) | 11 | 1
Statistical Analysis 1: Comparison: Self-directed Care vs Services as Usual; This mixed effects random regression analysis tested whether intervention participants would report greater likelihood of enrollment in educational classes that would be maintained longitudinally; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 4.14, 95% CI 2-sided [1.50 to 11.44]

7. Secondary Outcome: Change in Mental Health Service Cost
Description: Mental health service cost is measured by the amount of reimbursement for a paid claim from the Texas Department of State Health Services Data Warehouse, It represents the amount of dollars paid for delivery of a discrete behavioral health service. Higher value = higher cost. Minimum = 1 and maximum = 5,493.
Time Frame: First 12 months of study participation; Second 12 months of study participation; total 24 months of study participation
Measure: Mean (Standard Deviation); unit: Dollar Amount
Arm/Group | Self-directed Care | Services as Usual
Number analyzed (Participants) | 114 | 102
Dollar Amount
  Diagnostic services: Year 1 | 36 (67) | 26 (54)
  Diagnostic services: Year 2 | 14 (43) | 14 (43)
  Psychotherapy: Year 1 | 229 (454) | 23 (118)
  Psychotherapy: Year 2 | 133 (346) | 12 (70)
  Skills Training: Year 1 | 4 (19) | 27 (71)
  Psychosocial Rehab: Year 1 | 311 (783) | 646 (1394)
  Psychosocial Rehab: Year 2 | 130 (421) | 177 (416)
  Case Management: Year 1 | 26 (165) | 31 (141)
  Case Management: Year 2 | 3 (15) | 39 (149)
  Peer Services: Year 1 | 11 (64) | 9 (41)
  Peer Services: Year 2 | 15 (101) | 13 (89)
  Inpatient Care: Year 1 | 223 (1270) | 344 (1405)
  Inpatient Care: Year 2 | 72 (476) | 269 (1385)
  Psychiatric Crisis Services:Year 1 | 121 (453) | 168 (407)
  Psychiatric Crisis Services: Year 2 | 70 (269) | 162 (574)
  Residential Support: Year 1 | 58 (336) | 23 (166)
  Residential Support: Year 2 | 58 (371) | 69 (386)
  Substance Abuse Treatment: Year 1 | 44 (227) | 203 (1029)
  Substance Abuse Treatment: Year 2 | 55 (385) | 90 (504)
  Medication Management: Year 1 | 182 (205) | 303 (229)
  Medication Management: Year 2 | 111 (162) | 200 (282)
  Medications: Year 1 | 1071 (2047) | 1387 (2574)
  Medications: Year 2 | 902 (2414) | 1218 (2993)
  Non-Traditional Services: Year 1 | 679 (516) | 0 (0)
  Non-Traditional Services: Year 2 | 667 (658) | 0 (0)
  Total Including Non-Traditional Services: Year 1 | 2998 (3128) | 3189 (4608)
  Total Including Non-Traditional Services: Year 2 | 2241 (2960) | 2303 (4266)
  Total Excluding Non-Traditional Services: Year 1 | 2319 (3316) | 3189 (4608)
  Total Excluding Non-Traditional Services: Year 2 | 1574 (2938) | 2303 (4266)

ADVERSE EVENTS:
Time Frame: The time frame over which adverse event data were collected was 3 years.
Description: For other serious adverse events, we included incarcerations.
Arm/Group | Self-directed Care | Services as Usual
All-Cause Mortality (participants affected / at risk) | 3/114 | 2/102
Serious Adverse Events (participants affected / at risk) | 1/114 | 0/102
Other Adverse Events (participants affected / at risk) | 12/114 | 11/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-directed Care (N=114) | Services as Usual (N=102)
Adverse events were monitored without regard to the specific adverse event term (Immune system disorders) | 1 (1) | 0 (0) — Subject was admitted to hospice care for HIV infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-directed Care (N=114) | Services as Usual (N=102)
Adverse events were monitored without regard to the specific adverse event term (Psychiatric disorders) | 0 (0) | 1 (1) — One participant became very upset and frustrated due to problems with mental health service provider (i.e., reported they violated her privacy and that she was treated disrespectfully).
Adverse events were monitored without regard to the specific adverse event term (Psychiatric disorders) | 12 (12) | 10 (10) — Incarceration of research subjects entirely unrelated to the research

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No